CLINICAL TRIAL: NCT01196793
Title: Evaluation of Medical and Non-medical Factors Associated With Admission of Children Aged 3 Months to 5 Years Presenting to the Urban Paediatric Emergency Department With Febrile Illness in the United Kingdom and in Switzerland
Brief Title: Hospital Admissions in Children Aged 3 Months to 5 Years Presenting With Fever to the Emergency Department
Status: Completed | Type: Observational
Sponsor: Imperial College Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: SMH 24062010 V1 4
Record Dates: First submitted 2010-09-06; First posted 2010-09-08 (Estimated); Results first posted 2019-09-09 (Actual); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: Fever
Keywords: Feverish illness in children
MeSH Terms: conditions — Fever

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- febrile children, age 3 m to 5 y

SUMMARY:
This study primarily aims to describe factors associated with hospitalisation of children aged 3 months to 5 years presenting with fever to an urban paediatric A&E departments by describing and analysing characteristics both of those patients admitted to hospital and those managed in the community. To complement this, information on the short-term healthcare utilization by families attending the emergency department because of feverish illness will be collected. The study will be carried out in one participating centre in Switzerland and the United Kingdom, respectively, to enable a head to head comparison of the assessment and admission practices in two European countries. The resulting data will be used as the basis for further research in this area and will provide information on how to optimally structure service provision in acute febrile childhood illness.

DETAILED DESCRIPTION:
A significant number of children 0 to 5 years of age are seen in paediatric Accident & Emergency departments (A&E) with feverish illness. Most of these patients could safely be managed in a primary care setting, particularly with guidelines in place on how to optimally assess these children. Some patients, however, will require admission, either because of a potentially serious underlying disease or because of other factors, for example parental concern or difficulties in communication because of language barriers. An increase in the number of children attending A&E departments with feverish illness as well as a rise in the volume of admissions has been noted over time. To enable an appropriate adaptation of acute medical services for children an in depth understanding of the assessment and admission processes is crucial.

ELIGIBILITY:
Inclusion Criteria:

* Child aged 3months to 5years
* Temperature above or equal to 38°C measured by any method or reported hot by parents

Exclusion Criteria:

* none

Ages: 3 Months to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children aged 3 months to 5 years presenting to an urban paediatric emergency department with fever
Sampling Method: Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2012-04-30 (Actual); Primary Completion 2014-07-03 (Actual); Study Completion 2014-07-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hermione Lyall, MD, Principal Investigator — Imperial College Healthcare NHS Trust
Locations (2):
- University Children's Hospital, Zurich, Switzerland
- St Mary's Hospital, Imperial NHS Hospitals Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Febrile Children, Age 3 m to 5 y: 3 month to 5 years old children with febrile illness
Period: Overall Study
Arm/Group | Febrile Children, Age 3 m to 5 y
Started | 108
Completed | 108
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Febrile Children, Age 3 m to 5 y
Number analyzed (Participants) | 108
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 108
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54
  Male | 54
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 108

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Admission to Hospital Due to Parental High Levels of Worry
Description: Interview with the patient family to evaluation of the reasons for admission to emergency department
Time Frame: 7-10 days
Measure: Count of Participants; unit: Participants
Groups:
- Febrile Children, Age 3 m to 5 y: 3 month to 5 years children with febrile
Arm/Group | Febrile Children, Age 3 m to 5 y
Number analyzed (Participants) | 108
Participants | 87

ADVERSE EVENTS:
Time Frame: 1 years
Groups:
- Febrile Children, Age 3 m to 5 y: 3 month to 5 years old children with febrile
Arm/Group | Febrile Children, Age 3 m to 5 y
All-Cause Mortality (participants affected / at risk) | 0/108
Serious Adverse Events (participants affected / at risk) | 0/108
Other Adverse Events (participants affected / at risk) | 0/108

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes